CLINICAL TRIAL: NCT01434966
Title: Changes in Quadriceps Function Following Local or Distant Interventions in Individuals With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCT11-16215
Record Dates: First submitted 2011-09-14; First posted 2011-09-15 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Patellofemoral Pain Syndrome; Chondromalacia Patellae; Anterior Knee Pain Syndrome
Keywords: Lumbopelvic Manipulation; Lumbosacral Manipulation; Sacroiliac Manipulation; TENS Spine; TENS Knee; Knee Pain; Chronic Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Chondromalacia Patellae | interventions — Transcutaneous Electric Nerve Stimulation; Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lumbopelvic Manipulation (Experimental): The lumbopelvic joint manipulation (Grade V mobilization) will be performed on the ipsilateral side of the test limb. The participant will be passively side-bent towards and rotated away from the selected lumbopelvic region which is followed by the delivery of a posterior/inferior force through the opposite anterior superior iliac spine. If a cavitation is not heard or felt by the patient or clinician, the technique will be repeated. If the second attempt does not produce cavitation the procedure will be repeated on the contralateral side using similar methods. If cavitation is not heard or felt by the participant or clinician following the second attempt on the contralateral side, the participant will proceed with the assessment of quadriceps strength and activation as usual.
  Interventions: Other: Lumbopelvic Manipulation
- TENS- Spine (Experimental): The TENS electrodes will be applied lateral to L1 and L2 and lateral to S5 and S1. The TENS unit will be set to deliver a continuous TENS biphasic pulsatile current at 150 Hz, with a phase duration of 150 microseconds. The TENS unit will be worn during all exercise testing and for the first 30 minutes of quadriceps force output and activation testing. After the 30 minute post-intervention measures (Post30) are obtained, the TENS unit will be turned off.
  Interventions: Other: TENS- Spine
- TENS- Knee (Experimental): The TENS electrodes will be applied on the medial and lateral superior, as well as the medial and lateral inferior, borders of the patella. Care will be taken not to place TENS electrodes on the quadriceps muscles or muscles of the anterior leg. The TENS unit will be set to deliver a continuous TENS biphasic pulsatile current at 150 Hz, with a phase duration of 150 microseconds. The TENS unit will be worn during all exercise testing and for the first 30 minutes of quadriceps force output and activation testing. After the 30 minute post-intervention measures (Post30) are obtained, the TENS unit will be turned off.
  Interventions: Other: TENS- Knee

INTERVENTIONS:
Other: Lumbopelvic Manipulation — The lumbopelvic joint manipulation (Grade V mobilization) will be performed on the ipsilateral side of the test limb. The participant will be passively side-bent towards and rotated away from the selected lumbopelvic region which is followed by the delivery of a posterior/inferior force through the opposite anterior superior iliac spine. If a cavitation is not heard or felt by the patient or clinician, the technique will be repeated. If the second attempt does not produce cavitation the procedure will be repeated on the contralateral side using similar methods. If cavitation is not heard or felt by the participant or clinician following the second attempt on the contralateral side, the participant will proceed with the assessment of quadriceps strength and activation as usual.
  Other Names: Grade V mobilization; High velocity, low amplitude thrust mobilization
  Arms: Lumbopelvic Manipulation
Other: TENS- Spine — The TENS electrodes will be applied lateral to L1 and L2 and lateral to S5 and S1. The TENS unit will be set to deliver a continuous TENS biphasic pulsatile current at 150 Hz, with a phase duration of 150 microseconds. The TENS unit will be worn during all exercise testing and for the first 30 minutes of quadriceps force output and activation testing. After the 30 minute post-intervention measures (Post30) are obtained, the TENS unit will be turned off.
  Other Names: Transcutaneous electrical nerve stimulation (TENS); Electrical stimulation
  Arms: TENS- Spine
Other: TENS- Knee — The TENS electrodes will be applied on the medial and lateral superior, as well as the medial and lateral inferior, borders of the patella. Care will be taken not to place TENS electrodes on the quadriceps muscles or muscles of the anterior leg. The TENS unit will be set to deliver a continuous TENS biphasic pulsatile current at 150 Hz, with a phase duration of 150 microseconds. The TENS unit will be worn during all exercise testing and for the first 30 minutes of quadriceps force output and activation testing. After the 30 minute post-intervention measures (Post30) are obtained, the TENS unit will be turned off.
  Other Names: Transcutaneous electrical nerve stimulation (TENS); Electrical stimulation
  Arms: TENS- Knee

SUMMARY:
The purpose of this study is to determine if interventions applied at a distant site, lumbopelvic region (manipulation and TENS), have a similar effect as interventions applied locally at the knee (TENS) on quadriceps force output and activation as well as reports of pain during common exercises in individuals with PFPS.

DETAILED DESCRIPTION:
Interventions for PFPS usually focus on strengthening the quadriceps muscle and hip musculature. It is suggest that intervention programs specifically address muscle inhibition beyond typical strengthening exercises. To specifically address decreased muscle activation transcutaneous electrical neuromuscular stimulation (TENS), applied to the knee, has been shown to reduce pain and increase muscle activation in individuals with knee osteoarthritis. Interventions including joint manipulation applied at distant sites, such as the lumbopelvic region have also been shown to increase muscle activation following intervention in individuals with PFPS, but the duration of effect is unknown. It is hypothesized that interventions which alter spinal afferent signals may have an effect on efferent motor output. Since the lumbopelvic region and the knee joint share common nerve root levels it is possible that interventions applied to either site may influence efferent motor output to the quadriceps muscle. The magnitude and duration of this effect is unknown.

Both TENS and lumbopelvic manipulation have also been shown to reduce pain during exercise in individuals with knee joint pathology. This study would better determine the magnitude of effective pain reduction between interventions applied at the knee joint and at a distant site, the lumbopelvic region.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-50 years
* Insidious onset of patellofemoral pain lasting greater than 1 month in duration
* Unilateral or Bilateral knee pain or dysfunction with at least two of the following symptoms: patella compression, squatting, prolonged sitting, going up or down stairs, or isometric quadriceps contraction.

Exclusion Criteria:

* Participants who are outside of age range (to ensure bony maturity while reducing the prevalence of age related degenerative changes and hypomobility.)
* Ligamentous insufficiency, meniscus damage, patellar tendonitis, history of subluxation/dislocation
* Participants with traumatic spine or lower extremity injury within past 6 months
* Participants who have had previous adverse reactions to electrical stimulation (i.e. electrode burns.)
* Participants with signs indicating lumbar nerve root compression or upper motor neuron lesions (contraindication for lumbopelvic joint manipulation)
* Participants with ankylosing spondylitis (contraindication for lumbopelvic manipulation)
* Participants with spinal cord disease or cauda equina (contraindication for lumbopelvic manipulation)
* Participants with osteoporosis (contraindication for lumbopelvic joint manipulation)
* Participants with rheumatoid arthritis (contraindication to lumbopelvic joint manipulation.)
* Participants who may be currently pregnant. (contraindication for electrical stimulation and lumbopelvic joint manipulation.)
* Participants who have a demand-type cardiac pacemaker (contraindication for electrical stimulation)
* Participants with diagnosis of cancer (current cancer is a contraindication for electrical stimulation and relative contraindication for lumbopelvic joint manipulation)
* Participants who are unable to give consent or are unable to understand procedures of experiment.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Quadriceps force output and activation | Single Study Visit
  Quadriceps activation will be estimated by utilizing the burst-superimposition technique on a maximum voluntary isometric contraction (MVIC) and during a resting condition. The burst-superimposition technique provides the muscle with a percutaneous stimulus to recruit any remaining muscle fibers which have not been stimulated.

SECONDARY OUTCOMES:
Knee pain during exercise | Single Study Visit
  Participants will perform three common exercises which include going up a step (20 cm), going down a step (20 cm) and squatting. Pain during activity will be assessed using a visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Grindstaff, PhD, PT, ATC, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States